CLINICAL TRIAL: NCT00709137
Title: Randomized Trial of Spironolactone Versus Amiloride as an Add on Agent in Resistant Hypertension
Brief Title: Spironolactone Versus Amiloride as an Add on Agent in Resistant Hypertension
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: VA Salt Lake City Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Richard Rose, Assistant Professor, VA Salt Lake City Health Care System
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB_00027466
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Hypertension
Keywords: resistant hypertensions; spironolactone; amiloride; ambulatory blood pressure monitoring
MeSH Terms: conditions — Hypertension | interventions — Spironolactone; Amiloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): this arm will include patients with resistant hypertension who are on 3 reasonably dosed agents (one being an appropriately dosed diuretic) and spironolactone will be added (dose range 12.5mg-50mg)
  Interventions: Drug: spironolactone
- 2 (Active Comparator): this arm will include patients with resistant hypertension who are on 3 reasonably dosed agents (one being an appropriately dosed diuretic) and amiloride will be added (dose range 2.5-10mg)
  Interventions: Drug: amiloride

INTERVENTIONS:
Drug: spironolactone — tablet form. doses used range from 12.5-50mg po QDAY. Total duration would be until completion or study or medication intolerance.
  Other Names: aldactone
  Arms: 1
Drug: amiloride — amiloride 2.5-10 mg po QDAY. Duration until completion of study or until tolerance
  Other Names: midamor
  Arms: 2

SUMMARY:
Joint National Committee 7 (JNC-7) defines resistant hypertension as a persistent elevation of blood pressure (BP) above goal - ≥ 140/90 mm Hg for the general hypertensive population or ≥ 130/80 mm Hg for persons with diabetes mellitus or chronic kidney disease - for at least three months despite treatment with three or more optimally dosed antihypertensive agents, including a diuretic. The exact prevalence of resistant hypertension is uncertain but may include 5-20% of hypertensive persons in primary care settings and 15-35% of the older, higher cardiovascular risk hypertensive patients incorporated into recent clinical trials of antihypertensive therapy. Observational studies demonstrate that patients with resistant hypertension experience a higher rate of cardiovascular and renal target organ damage such as left ventricular hypertrophy, microalbuminuria, and renal insufficiency and more cardiovascular disease (CVD) events than patients whose hypertension is well-controlled. Additionally, resistant hypertension patients may be subjected to the considerable expense of multiple office visits, diagnostic testing for secondary causes of hypertension, and referral to hypertension specialists. Because multiple factors can contribute to resistant hypertension, an explicit, sequential approach to evaluation and management is essential to optimize blood pressure, reduce cardiorenal morbidity and mortality, and avoid unnecessary expense. A number of observational studies have suggested the potential efficacy of both spironolactone and amiloride when added to a 3 drug antihypertensive regimen, but to date no randomized study has directly compared the two agents. The goal of this study is to determine whether spironolactone or amiloride is the more effective fourth agent to add to a three drug regimen in patients with resistant hypertension.

DETAILED DESCRIPTION:
m/a

ELIGIBILITY:
Inclusion Criteria:

* Participants will be selected from a broad range of medical clinics at the Salt Lake City VA Medical Center and surrounding community based outpatient clinics (CBOCs).
* The participants will be referred to a resistant hypertension clinic by either their primary care provider or by a subspecialist. The referrals are made via a computerized system that is used in the Veterans Affairs Medical Center (VA) called Computerized Patient Record System (CPRS).
* Patients are referred if their blood pressure is above goal as defined by JNC 7 and they are on 3 antihypertensive medications with one of the agents being a diuretic.
* All patients age 18 -80 years old.

Exclusion Criteria:

* Patients that will be excluded from the study if they have had a documented adverse reaction to either spironolactone or amiloride.
* diagnosis of primary hyperaldosteronism
* inability to adhere to frequent laboratory monitoring
* estimated glomerular filtration rate (GFR) < 45 ml/min/1.73m2
* baseline serum potassium above 5.0 mEq/L
* type 4 renal tubular acidosis
* pregnancy
* heart failure that meets criteria for using either eplerenone or spironolactone
* current unstable renal function

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-10; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Dose titration of spironolactone and amiloride will cease once the ABPM study reveals a goal 24 hour mean BP below 130/80 in the general hypertensive patients or below 120/70 in patients with diabetes mellitus or chronic kidney disease (eGFR < 60) | 2-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Rose, MD, Principal Investigator — Univ of Utah Division of General Internal Medicine; VAMC SLC Internal Medicine
Locations (1):
- VAMC SLC - George Wahlen VA, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Calhoun DA, Jones D, Textor S, Goff DC, Murphy TP, Toto RD, White A, Cushman WC, White W, Sica D, Ferdinand K, Giles TD, Falkner B, Carey RM; American Heart Association Professional Education Committee. Resistant hypertension: diagnosis, evaluation, and treatment: a scientific statement from the American Heart Association Professional Education Committee of the Council for High Blood Pressure Research. Circulation. 2008 Jun 24;117(25):e510-26. doi: 10.1161/CIRCULATIONAHA.108.189141. PMID 18574054
- [Background] Moser M, Setaro JF. Clinical practice. Resistant or difficult-to-control hypertension. N Engl J Med. 2006 Jul 27;355(4):385-92. doi: 10.1056/NEJMcp041698. No abstract available. PMID 16870917
- [Background] Nishizaka MK, Zaman MA, Calhoun DA. Efficacy of low-dose spironolactone in subjects with resistant hypertension. Am J Hypertens. 2003 Nov;16(11 Pt 1):925-30. doi: 10.1016/s0895-7061(03)01032-x. PMID 14573330
- [Background] Lane DA, Shah S, Beevers DG. Low-dose spironolactone in the management of resistant hypertension: a surveillance study. J Hypertens. 2007 Apr;25(4):891-4. doi: 10.1097/HJH.0b013e328014954d. PMID 17351384
- [Background] Lane DA, Beevers DG. Amiloride 10 mg is less effective than spironolactone 25 mg in patients with hypertension resistant to a multidrug regime including an angiotensin-blocking agent. J Hypertens. 2007 Dec;25(12):2515-6. doi: 10.1097/HJH.0b013e3282f254d9. No abstract available. PMID 17984678